CLINICAL TRIAL: NCT07397806
Title: Home-Based Leg Dexterity Trainer for Management of Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Steadman Philippon Research Institute (Other)
Collaborators: Neuromuscular Dynamics (Unknown); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Scott Tashman, Director, Biomedical Engineering, Steadman Philippon Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMD-OA-2024; R44AG090114 (NIH)
Record Dates: First submitted 2026-01-26; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Osteo Arthritis of the Knee
Keywords: osteoarthritis; knee; exercise; dexterity
MeSH Terms: conditions — Osteoarthritis; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Leg Dexterity Training (Experimental): For the Lex Dexterity Training group, participants will be seated at the edge of a standard-height (76 cm) table and instructed to hold on to the edge of the table and support their weight equally through the table and the support leg before placing the foot of the training leg on the device's platform. The training leg will be positioned in a standardized posture (85 - 95° of hip and knee flexion) with the foot on the platform. Participants will press down on the platform ten (10) times, one leg at a time. Subjects will be asked to reach and hold the maximal force they can sustain before the device becomes unstable, thus engaging and training their neuromuscular control of unstable foot-ground interactions. After the initial in-person training session, participants will take the device home, with instructions to complete the training protocol (approximately 10-minute sessions) 3 times per week. The sessions are guided and logged with a tablet-based app.
  Interventions: Device: Lex Dexterity Trainer
- Wobble Board (Active Comparator): The Wobble Board (Control) group will train for 10 minute sessions 3 times per week on a commercially available wobble board, with a safety rail system to provide support and prevent falls. The wobbleboard is a well-known, safe and moderately effective intervention for treating knee OA. This training will consist of 5 repetitions each of: (i) forward/backward and (ii) side-to-side board tilts, and 30 seconds of (iv) single-leg stance on each leg. As previously described, this wobbleboard protocol is a safe and effective intervention in knee OA. As shown, the wobble board is equipped with safety bars to protect against falls. After the initial in-person training session, participants will take the wobble board and safety rails home, with instructions to complete the training protocol (approximately 10-minute sessions) 3 times per week. The sessions are guided and logged with a tablet-based app.
  Interventions: Device: Wobble Board

INTERVENTIONS:
Device: Lex Dexterity Trainer — The Leg Dexterity Trainer is a portable, wireless device. A seated participant uses their foot to compress a platform atop a slender spring, which becomes unstable as it begins to buckle at low forces. The participant must then control their leg dexterity (i.e., via short-latency sensorimotor circuits) to stabilize the unstable dynamic foot-ground interactions.
  Arms: Leg Dexterity Training
Device: Wobble Board — A wobble board is a circular or rectangular board with a rounded base, designed to improve balance, core strength, and coordination by creating an unstable surface that challenges stability.
  Arms: Wobble Board

SUMMARY:
Rationale:

Roughly 14 million adults aged 60 or older (10% male/13% female) in the United States experience symptoms of knee osteoarthritis (OA). Knee OA pain progressively impacts aging, reducing mobility and increasing morbidity. Nonsurgical self-management of knee OA includes exercise to promote proper knee mechanics, non-steroidal anti-inflammatory drugs (NSAIDs), cortisone injections, and weight loss to reduce pain and retain function. As OA has no cure, self-management progresses to ~1 million joint replacements per year. Critically, home-based devices are lacking for specifically training the low-level proprioceptive and neuromuscular circuitry for proper knee mechanics in a safe, focused, mechanistic way. Such devices would supplement exercises for strength, mobility, and whole-body loading and movement.

Initially considered a wear-and-tear condition, knee OA is now understood as a complex disease involving inflammatory responses to mechanical loading and neuromuscular feedback loops among pain, joint damage, and dynamic loading. Home-based exercises remain a primary nonpharmacological and nonsurgical approach to managing chronic pain in OA that fundamentally disrupts proprioception and neuromuscular control of the joint, which accelerates articular degeneration.

Neuromuscular Dynamics, LLC has developed a simple, safe, quick, and effective Leg Dexterity System that is portable, wireless, and coupled to HIPAA-compliant cloud analytics. A seated participant uses their foot to compress a platform atop a slender spring, which becomes unstable as it begins to buckle at low forces. The participant must then control their leg dexterity (i.e., via short-latency sensorimotor circuits) to stabilize the unstable dynamic foot-ground interactions. A tablet computer connected to the device provides feedback during use and uploads the participant's activity data to the server for analysis and reporting, accessible to users and clinicians.

The investigators have successfully tested Leg Dexterity in control participants in multiple publications. The Leg Dexterity test is safe and poses minimal risk as the forces needed to do it are very low, does not involve full weight- bearing maneuvers, and is performed while seated without the risk of falling.

Study:

The investigators will conduct a randomized home-based clinical trial in knee OA to demonstrate the efficacy of leg dexterity training to reduce pain and improve function compared to currently prescribed dynamic exercise on a wobble board (a commonly used approach for improving proprioception and balance). Successful completion of this study will justify the adoption of the Leg Dexterity System as an effective at-home supplement to any nonsurgical management of knee OA.

The investigators propose a longitudinal double-blind dose-matched trial comparing 8 weeks of leg dexterity training (Treatment using a slender, unstable spring system that engages short-latency sensorimotor control, 42 participants) vs. at-home wobble board exercises (Control, 42 participants) at the Steadman Philippon Research Institute.

DETAILED DESCRIPTION:
The investigators will conduct a randomized home-based clinical trial in knee OA to demonstrate the efficacy of leg dexterity training to reduce pain and improve function compared to currently prescribed dynamic exercise on a wobble board (a commonly used approach for improving proprioception and balance). Successful completion of this study will justify the adoption of the Leg Dexterity System as an effective at-home supplement to any nonsurgical management of knee OA.

The investigators propose a longitudinal double-blind dose-matched trial comparing 8 weeks of leg dexterity training (Treatment using a slender, unstable spring system that engages short-latency sensorimotor control, 42 participants) vs. at-home wobble board exercises (Control, 42 participants) at the Steadman Philippon Research Institute.

Primary Hypothesis: Neuromuscular control: Compared to the Control group, the Treatment group will report greater reduction in knee pain and demonstrate improved function in the more-affected leg. The primary outcomes measures will include The Western Ontario and McMaster Universities Arthritis Index (WOMAC) Pain subscale and the Single Limb Stance Test (SLS).

Secondary Hypothesis: Whole-body function: Compared to the Control group, greater OA-related whole-body functional improvements will be found in the Treatment group. Secondary outcome measures include the WOMAC stiffness and physical function subscales; International Knee Documentation Committee (IKDC) Subjective Knee score, Timed-up-and-go test (TUG); 6 min walk test (6MW); 40-meter walk (40mW) Test; and lower-extremity Gait analysis.

The Leg Dexterity System:

To use the Leg Dexterity system, seated individuals are instructed to use a single leg to slowly compress the spring with the platform with the goal to make the force feedback line as high as possible (i.e., maximize vertical compression force) throughout each ~10 second trial without letting the foot slip on the platform (see Figure). The spring begins to show instabilities at low forces. Participants are informed that it is ok for the spring to bend and oscillate (i.e., due to the instability inherent in task). Despite the motion, the goal is to maintain the highest possible force level without the spring buckling (which occurs when the force exceeds 15% of body weight). Because the spring becomes increasingly instable even at these low forces, the maximal sustained compression quantifies their maximal neuromuscular control abilities.

The Wobble Board:

Commercial wobble boards (Core-Tex Reactive Trainer, Core-Tex Fitness, Inc. shown at right). are an intervention used at home and the clinic to improve leg and body dynamic control. As shown, the wobble board is equipped with safety bars to protect against falls and poses minimal risk for older adults and adults with knee OA. To use the wobble board with eyes open, participants will stand on the center of the board and perform 5 repetitions each of: (i) forward/backward and (ii) side-to-side board tilts, and 30 seconds of (iv) single-leg stance on each leg. This wobbleboard protocol is a safe and effective intervention in knee OA[67,68], and participants are encouraged to minimize the use of the handle bars within their comfort level to maximize and improve leg and body dynamic control.

Participant Assignment:

After informed consent, study participants will undergo a baseline assessment and be randomized to receive either the Leg Dexterity device or the wobbleboard. They will then take their assigned device home, with instructions to perform the exercises they were trained on 3 times per week for 8 weeks and maintain a log of their activities. After 8 weeks, they will return to the Steadman Philippon Research Institute for a repeat assessment and to return the equipment.

Establish the clinical feasibility, utility and efficacy of using a home-based Leg Dexterity training program to reduce pain and improve function for individuals with osteoarthritis.

There is a single endpoint at 8 weeks after initiation of training.

• 82 patient participants with knee osteoarthritis, targeting equal numbers of male and female participants.

This is a Phase II clinical trial, providing an initial assessment of efficacy.

Single-center study conducted at the Steadman Philippon Research Institute in Vail, CO

Participants will be randomized into one of two home treatment regimens, utilizing either the Leg Dexterity system or a commercially available wobbleboard. Training will occur 3 times per week for 8 weeks.

36 months

The initial visit will consist of informed consent, screening, baseline testing and training on the proper use of either the Knee Dexterity system or the wobbleboard. This visit will take approximately 3 hours. Participants will then conduct 8 weeks of home-based training using their assigned device. They will then return for their follow-up visit, during which the assessments performed at baseline will be repeated. This visit will take approximately 90 minutes. The supplied training device will be returned and study participation will be complete. Total study duration for each participant will be approximately 10 weeks.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Age 40 to 85 years
2. Ambulatory in home and community settings
3. History of knee osteoarthritis in one or both knees (Kellgren-Lawrence grade II-IV)
4. Baseline pain of 3-10 points on the target (i.e., more-affected) knee and a pain differential of at least -2 points on the contralateral knee as exhibited by the worst pain score for the previous week (on the 11-point Numeric Rating Scale, NRS/Visual Analog Scale VAS).
5. Capacity to personally give informed consent (consent via a legally authorized representative will not be accepted) and who are willing to comply with all study-related procedures and assessments

EXCLUSION CRITERIA:

1. Previous or Planned Knee Surgeries, Procedures, and/or Treatments:

   1. Planned surgery on either the contralateral or target knee at any time during the Study period, including pre-and post-training assessments.
   2. Within 6 months of signing informed consent has received diagnostic arthroscopy of the target knee or arthroscopic surgery (including microfracture and meniscectomy) on the target knee;
   3. Within 12 weeks of signing informed consent has received intra-articular treatment of the target knee with steroids or hyaluronic acid derivatives;
   4. Planned intra-articular treatment of the target knee with steroids or hyaluronic acid derivatives on either the contralateral or target knee at any time during the Study period including pre-and post-training assessments.
   5. History of previous total or partial arthroplasty in the target knee. Partial or total arthroplasty in the contralateral knee is acceptable as long as the surgery was performed at least 6 months prior to enrollment and the operative knee is asymptomatic
2. Current and/or Previous Medical Conditions, Surgeries, and/or Procedures:

   1. Within 2 years of signing informed consent, history of active blood disorders (i.e., DVTs, chronic blood clotting, hemophilia, leukemia, myeloma, etc.); or active malignancy of any type or history of a malignancy (with the exception of subjects with a history of treated basal or squamous cell carcinoma).
   2. Current diagnosis of fibromyalgia based on American College of Rheumatology (ACR) criteria.
   3. Any active known or suspected systemic autoimmune disease (except for vitiligo, residual auto-immune hypothyroidism requiring hormone replacement only, psoriasis not requiring systemic treatment for two years, conditions not expected to recur in the absence of an external trigger) or any history of systemic inflammatory arthritis such as psoriatic, rheumatoid, ankylosing spondylitis or reactive arthritis.
   4. Current or prior history of other joint diseases including but not limited to joint dysplasia, crystal-induced arthropathy (such as gout, or calcium pyrophosphate deposition disease evidenced by clinical and/or radiographic means), aseptic osteonecrosis, acromegaly, Paget's disease, Ehlers-Danlos Syndrome, Gaucher's disease, Stickler syndrome, joint infection, hemochromatosis, or neuropathic arthropathy of any cause.
   5. Any medical condition, including findings in laboratory or medical history or in the baseline assessments, that (in the opinion of the Principal Investigator or his designee) constitutes a risk or contraindication for participation in the Study or that could interfere with the Study conduct, endpoint evaluation or prevent the subject from fully participating in all aspects of the Study.
3. Within 8 weeks of signing informed consent, has used opioid analgesics and is not willing to discontinue these medications through the duration of the study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain: Numerical Rating Scale | Pain will be assessed during the baseline visit and after the 8-week training session.
  Study participants will complete the 11-point Numerical Rating Scale (NRS), which is a simple and frequently used pain assessment tool across both clinical research and clinical practice. The resulting score is a unitless integer ranging from 0 to 10, with 0 being no pain and 10 being the most pain imaginable.
Pain and Function: WOMAC | Womac will be assessed during the baseline visit and after the 8-week training session.
  Study participants will complete the Western Ontario McMaster Osteoarthritis Index (WOMAC) pain subscale, which consists of 5 questions about pain experienced during activities like walking, using stairs, and standing. Each item is rated on a 5-point Likert scale from 0 to 4: 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = extreme. Scores from each subsale are summed to produce a unitless pain/function score.

SECONDARY OUTCOMES:
Single Leg Stance Test: stance time | Baseline and after completion of the 8-week training session
  During the SLS, participants will be asked to maintain balance on each leg with their arms folded across their chest and eyes closed for at most 30 seconds on both stable (rigid surface) and unstable (e.g., 10 cm thick foam) surfaces on top of two Bertec® force plates with standardized software for SLS (Bertec, Inc., Columbus, OH). Participants will stand on the force plate and lift one foot off the floor (flexing the knee to approximately 60º) at their own pace and balance for up to 30 seconds. Trials will be terminated early upon ground contact with the non-test limb. Participants will complete three repetitions in each condition with each leg (12 total trials, 30 minutes for both legs). The first SLS outcome measure will be stance time.
Performance-Based Physical Function | Baseline and after completion of the 8-week training session
  Measures of functional performance will include the 6-minute walk test (6MW), timed-up-and-go test (TUG), and 4-meter walk (4mW) tests. The 6MW test measures the distance walked in 6 minutes to evaluate endurance. The TUG measures the time it takes a patient to rise from an armchair (seat height of 46 cm), walk 3 m, turn, and return to sitting in the same chair without physical assistance. The 4mW will be assessed at the fastest safe speed for each participant and assess the capacity for performance of certain activities (e.g., crossing a street before the light changes). These tests have been established as meaningful outcome measures in older persons with a wide range of conditions and have demonstrated validity and reliability.
Gait Analysis | Baseline and after completion of the 8-week training session
  Gait kinematics will be assessed using an 8-camera markerless motion capture system (Dari/Captury) during open-ground, free-speed walking. Three walking trials will be collected, with a minimum of 3 gait cycles per trial. Primary outcomes will be knee flexion angle (min/max/range and side-to-side symmetry) and stride parameters.
o 12-Item Short Form Health Survey (SF-12) | Baseline and after the 8-week training intervention
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life.
Single Leg Stance (SLS) test: Center of Mass Displacement | Baseline and after completion of the 8-week training session
  During the SLS, participants will be asked to maintain balance on each leg with their arms folded across their chest and eyes closed for at most 30 seconds on both stable (rigid surface) and unstable (e.g., 10 cm thick foam) surfaces on top of two Bertec® force plates with standardized software for SLS (Bertec, Inc., Columbus, OH). Participants will stand on the force plate and lift one foot off the floor (flexing the knee to approximately 60º) at their own pace and balance for up to 30 seconds. Trials will be terminated early upon ground contact with the non-test limb. Participants will complete three repetitions in each condition with each leg (12 total trials, 30 minutes for both legs). The second SLS outcome measure will be the mean and maximum displacement of the Center of Pressure (COP) location in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Tashman, PhD, Principal Investigator — Steadman Philippon Research Institute
Locations (1):
- Steadman Philippon Research Institute, Vail, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the reported results, after deidentification
Supporting Information: Study Protocol
Time Frame: IPD will be made available after publication of the final study results, for a period of 5 years.
Access Criteria: IPD will be available to Researchers who provide a methodologically sound proposal, by request to the study PI . To gain access, data requestors will need to sign a data access agreement.